CLINICAL TRIAL: NCT06810245
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Crossover Multicenter Study to Explore the Safety and Efficacy of Oral PIPE-791 as Treatment in Subjects With Chronic Osteoarthritis Pain (COAP) or Chronic Low Back Pain (CLBP)
Brief Title: Study of PIPE-791 for Subjects With Chronic Osteoarthritis Pain or Chronic Low Back Pain
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Contineum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTX-791-103
Record Dates: First submitted 2025-01-22; First posted 2025-02-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Chronic Osteoarthritis Pain; Chronic Low Back Pain
Keywords: chronic pain; pain; low back pain; osteoarthritis pain; osteoarthritis; pain management; neuropathic pain; CLBP; COAP; OA
MeSH Terms: conditions — Chronic Pain; Pain; Low Back Pain; Osteoarthritis; Agnosia; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active followed by Placebo (Experimental)
  Interventions: Drug: PIPE-791; Drug: Placebo
- Placebo followed by Active (Experimental)
  Interventions: Drug: PIPE-791; Drug: Placebo

INTERVENTIONS:
Drug: PIPE-791 — PIPE-791 tablet, taken once daily for 4 weeks
Drug: Placebo — Placebo tablet, taken once daily for 4 weeks

SUMMARY:
The primary goal of this clinical trial is to learn if PIPE-791 is safe and well-tolerated in adults with chronic osteoarthritis pain (COAP) or chronic low back pain (CLBP). The study will also explore whether PIPE-791 lowers pain in people with COAP or CLBP.

Subjects will:

* Complete a washout period to stop their current pain medications.
* Take a daily dose of PIPE-791 or placebo for 4 weeks, then reverse treatment assignment for another 4 weeks.
* Record pain levels and track dosing in a daily e-diary.
* Visit the clinic for checkups and lab tests throughout the study.
* Complete phone assessments during the treatment periods.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, 2-period crossover study designed to evaluate the safety and tolerability of PIPE-791 in approximately 20 adults with COAP and 20 adults with CLBP (with or without painful lumbosacral radiculopathy). Subjects will be randomized to receive either PIPE-791 or placebo daily for 4 weeks, followed by a crossover to the alternate treatment assignment for an additional 4 weeks.

A washout period of all chronic pain medications is required prior to randomization. Rescue medications, including acetaminophen and naproxen, will be permitted during the study.

Subjects will complete regular clinic visits for safety assessments, laboratory testing, and physical evaluations. Daily pain scores and dosing information will be reported by subjects using an electronic diary (e-diary).

All subjects who complete dosing will have a post-treatment safety follow-up/end of study (EOS) phone visit approximately 28 days after the last dose of study drug. Subjects who prematurely discontinue dosing and all assessments from the study will have an early termination (ET) visit as soon as possible on or after their last dose of study drug.

The total duration of participation, including screening, treatment, and follow-up, is approximately 16 weeks.

ELIGIBILITY:
Key Inclusion Criteria

* Male or female 18 to 70 years of age, inclusive, at the first Screening visit.
* Only one of the following chronic pain diagnoses at least 6 months prior to Screening:
* Osteoarthritis of the knee OR low back pain (with or without painful lumbosacral radiculopathy)
* Plain radiographs of the knee or lumbar spine consistent with diagnosis within 9 months prior to or during Screening.
* History of related daily pain for at least 6 months prior to Screening.
* Have a body mass index <40 (inclusive) at Screening.
* Willing to maintain a consistent regimen of any ongoing (stable format and frequency for the duration of study participation) non-pharmacologic pain-relieving therapies.
* Willing to discontinue medications taken for chronic pain conditions and usage of transcutaneous electrical nerve stimulation for the duration of the study.
* Male or female subjects with reproductive potential agree to comply with a highly effective contraceptive method as per protocol through 90 days after last study drug administration.
* Subjects taking systemic hormone-replacement therapy must be on a stable dose and regimen for at least 1 month prior to Screening.
* General good medical health with no clinically significant or relevant abnormalities except those attributed to the underlying chronic pain condition, including medical history, physical exam, vital signs, ECG, and laboratory evaluations (hematology, chemistry, and urinalysis) as assessed by the Investigator.
* Ability to use an eDiary to record daily pain scores.

Key Exclusion Criteria

* History of refractory chronic pain after multiple failed treatments as determined by the Investigator (e.g., no response to all of the following: surgery and/or nerve blocks, a regimen of at least two non-opioid pharmacotherapies, and physical rehabilitation, and weak opioids).
* Concurrent diagnosis of fibromyalgia or evidence of chronic widespread pain, or other pain that may interfere with the assessment of CLBP or COAP.
* Demonstrated noncompliance recording daily Numerical Rating Scale (NRS) scores during Screening.
* Have had a procedure within the past 6 months intended to produce permanent sensory loss in the target area of interest, e.g., an ablation procedure.
* Received capsaicin treatment (e.g., Qutenza) within the past 3 months prior to screening.
* Have surgery planned during the study for any reason, related or not, to the disease state under evaluation.
* Are non-ambulatory (use of assistive devices is allowed).
* History of Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, sarcoidosis, or amyloidosis.
* Diagnosed with OA during childhood or adolescence, including post-traumatic OA or OA due to genetic (e.g., hip dysplasia) or congenital (e.g., metabolic disorders) conditions.
* History of or clinical signs or symptoms of active joint infection, crystal disease of the knee, or a history of arthritis due to crystals (e.g., gout, pseudo gout).
* History of prior lumbar or thoracic spine surgery (e.g., discectomies, laminectomies, foraminotomies, or fusion).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Treatment-emergent adverse events (TEAEs) | For Treatment Period 1, from Baseline (Day 1) to End of Treatment Period 1 (TP1; Day 29), for Treatment Period 2, from Baseline of Treatment Period 2 (TP2; Day 29) to End of TP2 (Day 57).
  The number of subjects with TEAEs will be summarized in each treatment arm and compared within each treatment period.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Arizona Research Center, Phoenix, Arizona
  - Drug Studies America, Marietta, Georgia
  - Drug Trials America, Hartsdale, New York
  - Altoona Center of Clinical Research, Duncansville, Pennsylvania
  - JBR Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No